CLINICAL TRIAL: NCT06385951
Title: An Immersive Virtual Reality Spatial Navigation Task as Potential Biomarker for the Early Detection of Alzheimer's Disease.
Brief Title: Spatial Navigation for the Early Detection of Alzheimer's Disease.
Acronym: ALLO-task
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Principal Investigator, Prof. Dr. Paul Boon, Prof. Dr., University Hospital, Ghent
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ONZ-2023-0323
Record Dates: First submitted 2024-04-03; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Mild Cognitive Impairment; Alzheimer Disease; Healthy Aging
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients (Other): Patients with mild cognitive impairment and mild Alzheimer's dementia
  Interventions: Diagnostic Test: Procedure for patients
- Healthy volunteers (Other): Healthy volunteers
  Interventions: Diagnostic Test: Procedure for healthy controls

INTERVENTIONS:
Diagnostic Test: Procedure for patients — We will screen patients who undergo an MRI and neuropsychological examination as part of their diagnostic workup. If inclusion and exclusion criteria are met, patients will be asked to undergo additional investigations (FDG-PET, lumbar puncture, tau and amyloid PET and the ALLO iVR task).
  Arms: Patients
Diagnostic Test: Procedure for healthy controls — Healthy controls will be asked to undergo a neuropsychological examination, the ALLO iVR task, an MRI, FDG-PET and tau-PET.
  Arms: Healthy volunteers

SUMMARY:
Alzheimer's Disease (AD) is the most common form of dementia and may contribute to 60-70 % of all cases. An early, accurate diagnosis of AD will become increasingly important with disease-modifying therapies. Different types of fluid and neuroimaging biomarkers are available for the early detection of AD. However, implementation of routine use of these biomarkers in clinical settings is held back due to the risk of overdiagnosis, increased cost and invasiveness of the assessment method. Therefore, novel biomarkers are needed beyond the amyloid and tau pathologies for the early diagnosis of AD. Neuropsychological paper and pencil tests can detect AD and discriminate between different clinical stages. Since medial temporal lobe structures, including the hippocampus and entorhinal cortex (EC), are involved in spatial navigation and degenerate in the earliest stages of AD, spatial navigation can be considered as an early cognitive biomarker of the disease. Nonetheless, the measurement of spatial navigation needs further improvement since the current paper and pencil tests lack ecological validity. Therefore, the test environment should be set up in immersive Virtual Reality (iVR). Dr. Andrea Castegnaro (Space and Memory Lab of University College of London) developed the Allocentric Spatial Update Task (ALLO task), which is an iVR task measuring egocentric and allocentric spatial abilities.

Therefore, the main objective of this study is to evaluate whether allocentric and egocentric spatial navigation, measured by the ALLO iVR task can be considered a cognitive biomarker for the early detection of AD. In addition, the investigators want to report on the neuronal correlates of both spatial navigation strategies.

Through the Department of Neurology of the University Hospital of Ghent, which has a large cognitive disorders clinic, patients with mild cognitive impairment and mild Alzheimer's dementia will be recruited. Participants will undergo standard clinical assessment, including a neuropsychological examination, Magnetic Resonance Imaging, a 18F-fluorodeoxyglucose PET and a Lumbar Puncture. In addition, participants will also be asked to undergo Tau PET imaging, Amyloid PET imaging and complete the ALLO iVR task. Healthy controls will also be recruited and have to undergo the same investigations, except for the amyloid PET and lumbar puncture.

DETAILED DESCRIPTION:
Alzheimer's Disease (AD) is the most common form of dementia and may contribute to 60-70 % of all cases. It can be presented as a spectrum of progressive cognitive decline, with early episodic memory impairment, followed by progressive deterioration of other cognitive functions such as praxis, visual processing and spatial navigation. An early, accurate diagnosis of AD will become increasingly important with disease-modifying therapies. Different types of fluid and neuroimaging biomarkers are available for the early detection of AD. However, implementation of routine use of these biomarkers in clinical settings is held back due to the risk of overdiagnosis, increased cost and invasiveness of the assessment method. Therefore, novel biomarkers are needed beyond the amyloid and tau pathologies for the early diagnosis of AD.

Neuropsychological paper and pencil tests can detect AD and discriminate between different clinical stages. Traditionally, early episodic memory impairment has been considered the most specific cognitive biomarker of early AD. However, since medial temporal lobe structures, including the hippocampus and entorhinal cortex (EC), are involved in spatial navigation and degenerate in the earliest stages of AD, spatial navigation can also be considered as an early cognitive biomarker of the disease. Nonetheless, the measurement of spatial navigation needs further improvement since the current paper and pencil tests lack ecological validity. Therefore, we should evolve to a more innovative way of spatial navigation assessment that is more in line with the real world and set up the test environment in immersive Virtual Reality (iVR). Dr. Andrea Castegnaro (Space and Memory Lab of University College of London) developed the Allocentric Spatial Update Task (ALLO task), which is an iVR task measuring egocentric and allocentric spatial abilities.

Therefore, the main objective of this study is to evaluate whether allocentric and egocentric spatial navigation, measured by the ALLO iVR task can be considered a cognitive biomarker for the early detection of AD. In addition, the investigators want to report on the neuronal correlates of both spatial navigation strategies.

Through the Department of Neurology of the University Hospital of Ghent, which has a large cognitive disorders clinic, patients with mild cognitive impairment and mild Alzheimer's dementia will be recruited. Participants will undergo standard clinical assessment, including a neuropsychological examination, Magnetic Resonance Imaging, a 18F-fluorodeoxyglucose PET and a Lumbar Puncture. In addition, participants will also be asked to undergo Tau PET imaging, Amyloid PET imaging and complete the ALLO iVR task. Healthy controls will also be recruited and have to undergo the same investigations, except for the amyloid PET and lumbar puncture.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a Mild Cognitive Impairment (MCI) due to Alzheimer's Disease (AD)
* Patients with a mild Alzheimer's Dementia
* Patients with MCI without a formal dementia diagnosis
* Healthy controls

Exclusion Criteria:

* Diabetes (only for healthy controls)
* Epilepsy
* Presence of extreme depressive symptoms (>11 on Geriatric depression scale or >20 on Beck depression inventory)
* Presence of extreme anxiety (>22 on Beck Anxiety Inventory)
* A major psychiatric of medical disorder
* Alcohol excess
* Moderate to severe white matter lesions on MRI (>2 Fazekas)
* Any visual of mobility impairment of such severity as to compromise the ability to undertake the iVR task.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-10-01 (Estimated)

PRIMARY OUTCOMES:
Spatial navigation abilities | 1 hour
  Spatial navigation abilities (egocentric and allocentric) will be measured by means of the ALLO iVR task.

SECONDARY OUTCOMES:
Medial Temporal Lobe atrophy | 20 minutes
  MRI
Amount and spreading of amyloid in the brain | 1 hour
  Amyloid PET
Amount and spreading of tau in the brain | 1 hour
  Tau-PET
Decreases in cerebral glucose metabolism in the brain | 1 hour
  FDG-PET
Cognitive functioning | 1.5 hours
  Neuropsychologische examination
amyloidB1-42 / 40 ratio, total tau and phosphorylated tau | 1 hour
  Lumbar puncture

CONTACTS AND LOCATIONS:
Overall Officials: Paul Boon, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Gent, Ghent, East-Flanders, Belgium